CLINICAL TRIAL: NCT02755974
Title: Relationship Between Patient Phenotypes and Exacerbations in Chronic Obstructive Pulmonary Disease.
Brief Title: The London COPD Exacerbation Cohort
Acronym: EXCEL_Cohort
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 14IC1925
Record Dates: First submitted 2016-04-13; First posted 2016-04-29 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Sputum, Urine, Bronchoscopy brushing and Lavage fluid, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The London COPD exacerbation (EXCEL) cohort builds on an established cohort started in 1995 and designed to study COPD exacerbations and their impact on health-status and disease progression.

DETAILED DESCRIPTION:
Our intentions are to phenotype Chronic Obstructive Pulmonary Disease (COPD) patients on the basis of factors that a related to (a) exacerbation frequency which will include (b) lung function to assess disease severity, (c) baseline therapy, (d) airway and systemic inflammatory markers, (e) health status, (f) gene expression, (g) airway bacterial and viral load and (h) co-morbidity including cardiovascular disease, diabetes and psychological disease, (i) psychological factors,(j) mortality, (k) nasal susceptibility to rhinovirus infection, (l) heart rate variability (m) exhaled hydrogen sulphide.

ELIGIBILITY:
Inclusion Criteria:

* Forced Expiratory Volume in 1 sec (FEV1)/Forced Vital Capacity (FVC) ratio of <0.70
* Able and willing to give informed and written consent

Exclusion Criteria:

* Patients with a history of asthma, bronchiectasis, carcinoma of the bronchus, or other significant respiratory disease were excluded.
* Patients on Immunosuppressive medications or with active cancer
* Long term steroid therapy
* Age <40 years at recruitment

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD who are generally seen in outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Annual exacerbation rate (number of exacerbations over a 12 month period) | 12 months
  Definition of an exacerbation
  * The presence of 2 new symptoms (one of which must be major) for 2 consecutive days
  * Major symptoms: increased breathlessness (A), increased sputum colour (B1) or increased sputum amount (B2)
  * Minor symptoms: a cold (C), increased wheeze or chest tightness (D), Sore throat (E1), Increased cough (E2), Fever (F)

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga Wedzicha, Principal Investigator — Imperial College London
Locations (1):
- National Heart and Lung Institute, Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No